CLINICAL TRIAL: NCT03247491
Title: Effectiveness of a Mindfulness and Compassion Group Intervention Applied to Pregnant Women and Their Partners to Decrease Stress, Negative Affect and Depression During Pregnancy and Breastfeeding. Controlled and Randomized Study
Brief Title: Effectiveness of a Mindfulness and Compassion Intervention for Pregnant Women and Their Partners for the Prevention of Stress and Depression During Pregnancy and Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Javier Garcia Campayo (Other)
Collaborators: Universidad Nacional de Educación a Distancia (Other)
Responsible Party: Sponsor-Investigator, Javier Garcia Campayo, Co-director of Olga Sacristán´s (principal investigator) ph dissertation, Hospital Miguel Servet
Organization: Hospital Miguel Servet (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 50/2014/04
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Pregnancy, Childbirth and Postpartum
Keywords: Mindfulness; Compassion; Depression during Pregnancy and Postpartum; Prevention; Stress
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): TAU + mindfulness applied face to face 8 sessions of 120 minutes/session Mindfulness and Compassion based intervention applied in groups of 12-15 people in traditional format. Written material and sound recordings will be offered as support elements. The estimated duration of the face to face program is two months.
  Interventions: Behavioral: Mindfulness
- No intervention (No Intervention): Usual medical treatment (TAU) In this group the midwife will apply the usual treatment (childbirth education class in the third trimester of pregnancy).

INTERVENTIONS:
Behavioral: Mindfulness — TAU + mindfulness applied face to face 8 sessions of 120 minutes/session Mindfulness and Compassion based intervention applied in groups of 12-15 people in traditional format. Written material and sound recordings will be offered as support elements. The estimated duration of the face to face program is two months.
  Arms: Experimental

SUMMARY:
The aim of this study is to assess a mindfulness and compassion group intervention for pregnant women and their partners (8 weeks) for the prevention, reduction and treatment of stress, negative affect and depression in pregnancy and breastfeeding. This group intervention will also be compared with a Treatment as usual (TAU) group consisting in a childbirth education class taught by the Health Center midwife. The principal hypothesis is that the mindfulness and compassion intervention will be more effective than TAU.

DETAILED DESCRIPTION:
The aim of this study is to assess a mindfulness and compassion group intervention for pregnant women and their partners (8 weeks) for the prevention, reduction and treatment of stress, negative affect and depression in pregnancy and breastfeeding.

There will be two groups:

1. A face to face mindfulness and compassion intervention for pregnant women in their second trimester of pregnancy and their partners in group format (8 weeks) based in the Mindfulness Based Childbirth and Parenting program from Nancy Bardacke. This group will also receive in their third trimester of pregnancy the childbirth education classes taught by midwives (6-8 weeks) that every pregnant woman normally attends to in the National Health Care System in Spain (TAU).
2. A control group that will receive only the childbirth education class by midwives (TAU) group consisting in a childbirth education class taught by the Health Center midwife at the third trimester of pregnancy.

Each group will be composed of 60 participants with a total sample of 120. The principal hypothesis is that the mindfulness and compassion intervention will be more effective than TAU in the decrease of stress, negative affect and depression and in the increase of positive affect during pregnancy and breastfeeding.

The differences between the intervention and control group will be analyzed. Finally, a qualitative study will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old
* Willingness to participate in the study and signing informed consent
* Ability to understand and write Spanish.
* Women will be in their 6 to 25 weeks of pregnancy.
* All women eligible will be accepted with our without their partner.

Exclusion Criteria:

* Any diagnose of disease that may affect central nervous system (brain pathology, traumatic brain injury, dementia, etc.),
* Other psychiatric diagnoses or acute psychiatric illness (substance dependence or abuse, history of schizophrenia or other psychotic disorders, eating disorders, etc.),
* Any medical, infectious or degenerative disease that may affect mood, presence of delusional ideas or hallucinations consistent or not with mood, and suicide risk
* Currently taking psychopharmacological medication or under psychopharmacological treatment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Edinburgh postnatal depression scale (EPDS) | Baseline
  In the mindfulness and compassion based intervention group
Edinburgh postnatal depression scale (EPDS) | Baseline
  In the TAU control group
Edinburgh postnatal depression scale (EPDS) | Post-treatment 8 weeks from baseline in intervention group
Edinburgh postnatal depression scale (EPDS) | Post-treatment 8 weeks from baseline in TAU control group
Edinburgh postnatal depression scale (EPDS) | Post-partum 3 months follow up in 8 weeks intervention group
Edinburgh postnatal depression scale (EPDS) | Post-partum 3 months follow up in TAU control group
Edinburgh postnatal depression scale (EPDS) | Post-partum 6 months follow up in 8 weeks intervention group
Edinburgh postnatal depression scale (EPDS) | Post-partum 6 months follow up in TAU control group

SECONDARY OUTCOMES:
Sociodemographic data Gender, age, marital status, education, occupation, economical level | Baseline
  In the mindfulness-based intervention applied face-to-face and TAU control group
M.I.N.I. International Neuropsychiatric Interview | baseline applied in TAU and in intervention group
  only if needed
Client service receipt inventory (CSRI) | Baseline
  In the mindfulness-based intervention applied face-to-face and TAU control group
Client service receipt inventory (CSRI) | Post-partum 6 months follow up in 8 weeks intervention group
Client service receipt inventory (CSRI) | Post-partum 6 months follow up in TAU control group
Medical data regarding delivery and breastfeeding | 2 months after delivery
  In the mindfulness-based intervention applied face-to-face and TAU control group
Perceived Stress Scale (PSS) | Baseline
  In the mindfulness and compassion based intervention group
Perceived Stress Scale (PSS) | Baseline
  In the TAU control group
Perceived Stress Scale (PSS) | Post-treatment 8 weeks from baseline in 8 weeks intervention group
Perceived Stress Scale (PSS) | Post-treatment 8 weeks from baseline in TAU control group
Perceived Stress Scale (PSS) | Post-partum 3 months follow up in 8 weeks intervention group
Perceived Stress Scale (PSS) | Post-partum 3 months follow up in TAU control group
Perceived Stress Scale (PSS) | Post-partum 6 months follow up in 8 weeks intervention group
Perceived Stress Scale (PSS) | Post-partum 6 weeks follow up in TAU control group
Positive and negative affect (PANAS) | Baseline
  In the mindfulness and compassion based intervention group
Positive and negative affect (PANAS) | Baseline
  In the TAU control group
Positive and negative affect (PANAS) | Post-treatment 8 weeks from baseline in 8 weeks intervention group
Positive and negative affect (PANAS) | Post-treatment 8 weeks from baseline in TAU control group
Positive and negative affect (PANAS) | Post-partum 3 months follow up in 8 weeks intervention group
Positive and negative affect (PANAS) | Post-partum 3 months follow up in TAU control group
Positive and negative affect (PANAS) | Post-partum 6 months follow up in 8 weeks intervention group
Positive and negative affect (PANAS) | Post-partum 6 months follow up in TAU control group
Five Facets and factors of mindfulness (FFMQ) | Baseline
  In the mindfulness and compassion based intervention group
Five Facets and factors of mindfulness (FFMQ) | Baseline
  In the TAU control group
Five Facets and factors of mindfulness (FFMQ) | Post-treatment 8 weeks from baseline in 8 weeks intervention group
Five Facets and factors of mindfulness (FFMQ) | Post-treatment 8 weeks from baseline in TAU control group
Five Facets and factors of mindfulness (FFMQ) | Post-partum 3 months follow up in 8 weeks intervention group
Five Facets and factors of mindfulness (FFMQ) | Post-partum 3 months follow up in TAU control group
Five Facets and factors of mindfulness (FFMQ) | Post-partum 6 months follow up in 8 weeks intervention group
Five Facets and factors of mindfulness (FFMQ) | Post-partum 6 months follow up in TAU control group
Self Compassion Scale (SCS) | Baseline
  In the mindfulness and compassion based intervention group
Self Compassion Scale (SCS) | Baseline
  In the TAU control group
Self Compassion Scale (SCS) | Post-treatment 8 weeks from baseline in 8 weeks intervention group
  In the mindfulness and compassion based intervention group
Self Compassion Scale (SCS) | Post-treatment 8 weeks from baseline in TAU control group
Self Compassion Scale (SCS) | Post-partum 3 months follow up in 8 weeks intervention group
Self Compassion Scale (SCS) | Post-partum 3 months follow up in TAU control group
Self Compassion Scale (SCS) | Post-partum 6 months follow up in 8 weeks intervention group
Self Compassion Scale(SCS) | Post-partum 6 months follow up in TAU control group
Parental Evaluation Scale (EEP) | Post-partum 3 months follow up in 8 weeks intervention group
Parental Evaluation Scale (EEP) | Post-partum 3 months follow up in TAU control group
Parental Evaluation Scale (EEP) | Post-partum 6 months follow up in 8 weeks intervention group
Parental Evaluation Scale (EEP) | Post-partum 6 months follow up in TAU control group

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Nacional de Educacion a Distancia, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duncan LG, Bardacke N. Mindfulness-Based Childbirth and Parenting Education: Promoting Family Mindfulness During the Perinatal Period. J Child Fam Stud. 2010 Apr;19(2):190-202. doi: 10.1007/s10826-009-9313-7. Epub 2009 Oct 10. PMID 20339571
- [Background] Duncan, L.G., Cohn, M.A., Chao, M.T., Cook, J.G., Riccobono, J., & Bardacke, N. (2014a) Mind in labor: Effects of mind/body training on childbirth appraisals and pain medication use during labor. The Journal of Alternative and Complementary Medicine, 20, A17-A17.
- [Background] Duncan, L.G., Cohn, M.A., Cook, J.G., Hecht, F.M., & Bardacke, N. (2014b) The mind in labor: Employing mindfulness to alleviate fear and pain in childbirth. Poster presented at the 2nd biennial International Symposium for Contemplative Studies. Boston, MA.
- [Background] Duncan LG, Shaddix C. Mindfulness-Based Childbirth and Parenting (MBCP): Innovation in Birth Preparation to Support Healthy, Happy Families. Int J Birth Parent Educ. 2015 Jan;2(2):30-33. No abstract available. PMID 29051821
- [Background] Duncan LG, Cohn MA, Chao MT, Cook JG, Riccobono J, Bardacke N. Benefits of preparing for childbirth with mindfulness training: a randomized controlled trial with active comparison. BMC Pregnancy Childbirth. 2017 May 12;17(1):140. doi: 10.1186/s12884-017-1319-3. PMID 28499376
- [Derived] Sacristan-Martin O, Santed MA, Garcia-Campayo J, Duncan LG, Bardacke N, Fernandez-Alonso C, Garcia-Sacristan G, Garcia-Sacristan D, Barcelo-Soler A, Montero-Marin J. A mindfulness and compassion-based program applied to pregnant women and their partners to decrease depression symptoms during pregnancy and postpartum: study protocol for a randomized controlled trial. Trials. 2019 Nov 28;20(1):654. doi: 10.1186/s13063-019-3739-z. PMID 31779683